CLINICAL TRIAL: NCT04302909
Title: The Effectiveness of Focused Extracorporeal Shock Wave Therapy in the Treatment of Carpal Tunnel Syndrome: A Pilot Study
Brief Title: Effectiveness of fESWT in the Treatment of CTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Richard Crevenna, Ao.Univ.-Prof. Dr., MMSc. MBA, Head of the Department of Physical Medicine, Rehabilitation and Occupational Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1080/2019
Record Dates: First submitted 2020-03-02; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: focused extracorporeal shock wave therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): fESWT
  Interventions: Other: focused extracorporeal shock wave therapy; Other: night splint
- Sham Comparator (Sham Comparator): Sham fESWT
  Interventions: Other: sham focused extracorporeal shock wave therapy; Other: night splint

INTERVENTIONS:
Other: focused extracorporeal shock wave therapy — 40 Patients with mild to moderate CTS will be randomized to receive either fESWT (1-session a week for 3 weeks) or sham fESWT(1-session a week for 3 weeks). All subjects will be asked to wear night splints.
  Arms: Active Comparator
Other: sham focused extracorporeal shock wave therapy — 40 Patients with mild to moderate CTS will be randomized to receive either fESWT (1-session a week for 3 weeks) or sham fESWT(1-session a week for 3 weeks). All subjects will be asked to wear night splints.
  Arms: Sham Comparator
Other: night splint — 40 Patients with mild to moderate CTS will be randomized to receive either fESWT (1-session a week for 3 weeks) or sham fESWT(1-session a week for 3 weeks). All subjects will be asked to wear night splints.

SUMMARY:
The carpal tunnel syndrome (CTS) is the most common entrapment neuropathy in the general population.The focus extracorporeal shock wave (fEWST) is a non invasive treatment for various diseases. FESWT is new and potential treatment for peripheral nerve entrapment/ peripheral neuropathy . But there is still little known about the effects and long term effects of fESWT in the treatment of CTS.

DETAILED DESCRIPTION:
The aim of this study is to determine the effectiveness of fESWT in patients with carpal tunnel syndrome compared to participants receiving only night splint. Therefore 40 patients with mild to moderate CTS (verified by nerve conduction velocity) will be randomized to receive either fESWT (1-session a week for 3 weeks) or sham fESWT(1-session a week for 3 weeks). All subjects will be asked to wear night splints.

Evaluation will be performed at baseline (VAS, hand grip, electrodiagnostic parameters, questionnaires), 3 weeks (VAS, hand grip, questionnaires), 12 and 24 weeks (VAS, hand grip, electrodiagnostic parameters, questionnaires) after treatment.

ELIGIBILITY:
Inclusion Criteria:

- mild to moderate CTS verified by nerve conduction velocity

Exclusion Criteria:

* metabolic diseases
* blood clotting problems
* systemic diseases
* polyneuropathy
* chemotherapy during the study
* corticosteroid therapy
* use of anticoagulation
* history of trauma/surgery or nerve lesion of the teated extremity
* CTS surgery on the affected hand
* ICD/ pacemaker implantation
* other therapy for the affected hand during the study
* acute inflammation or infections
* severe mental illnesses/psychiatric diseases
* severe neurological diseases

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
VAS | baseline, 3th,12th and 24th weeks after treatment
  Visual Analog Scale: Change from baseline of pain 3th,12th and 24th weeks after treatment.

SECONDARY OUTCOMES:
hand grip strength | baseline, 3th,12th and 24th weeks after treatment
  hand grip strength:
distal motor latency of the median nerve | baseline,12th and 24th weeks after treatment
  electrophysiological parameter, using nerve conduction velocity to measure distal motor latency and antidromic sensory nerve conduction velocity of the median nerve.
  Change from baseline in conduction velocity of median nerve on 12th and 24th weeks after treatment.
sensory conduction velocity of the median nerve | baseline, 12th and 24th weeks after treatment
  electrophysiological parameter, using nerve conduction velocity to measure distal motor latency and antidromic sensory nerve conduction velocity of the median nerve.
  Change from baseline in conduction velocity of median nerve on 12th and 24th weeks after treatment.
SF-36 | baseline, 3th,12th and 24th weeks after treatment
  36-item Short Form Health Survey: Change from baseline in quality of life 3th,12th and 24th weeks after treatment.
Boston Scale | baseline, 3th,12th and 24th weeks after treatment
  Boston Symptom Severity Score: Change from baseline in severity of symptoms and functional status 3th,12th and 24th weeks after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Crevenna, Ao.Univ.-Prof. Dr., MMSc, MBA, Principal Investigator — Medical University of Vienna, Department of Physical Medicine, Rehabilitation and Occupational Medicine
Locations (1):
- Medical University of Vienna, Department of Physical Medicine, Rehabilitation and Occupational Medicine, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No